CLINICAL TRIAL: NCT00819533
Title: A Prospective, Open-Label, Single-Arm, Single-Center Study Evaluating the Preliminary Safety and Accuracy of the ActiSight Needle Guidance System in Patients Undergoing CT-Guided Percutaneous Chest Aspiration and Biopsy
Brief Title: Safety & Accuracy Study of the ActiSight Needle Guidance System in Patients Undergoing CT-Guided Percutaneous Chest Aspiration and Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ActiViews Ltd. (Industry)
Responsible Party: Uri Shreter, PhD / Study Director, ActiViews
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ASNG-LFNA-101-CAN
Record Dates: First submitted 2009-01-08; First posted 2009-01-09 (Estimated); Last update posted 2009-12-29 (Estimated); Status verified 2009-12

CONDITIONS: Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- sensor (Experimental): Patients will have their lung sample obtained under CT and ActiSight needle guidance system
  Interventions: Device: sensor (ActiSight™ Needle Guidance System)

INTERVENTIONS:
Device: sensor (ActiSight™ Needle Guidance System) — Patients will have their lung sample obtained under CT and ActiSight needle guidance system

SUMMARY:
This study is designed to evaluate preliminary safety and accuracy of the ActiSight™ Needle Guidance System in patients undergoing CT-guided lung aspiration or biopsy. This image guidance system uses a combination of CT scans and camera images to help guide a biopsy needle to a lung lesion. The system displays a simulated image of a biopsy needle and its estimated path for the biopsy.

DETAILED DESCRIPTION:
Why is this study conducted to demonstrate the safety and effectiveness of the ActiSight Needle Guidance System in assisting trained physicians perform CT guided percutaneous needle biopsy (PNB) and fine needle aspiration (FNA) procedures in the chest.

Subjects, who are scheduled for medically indicated chest PNB or FNA procedures and meet all the inclusion and exclusion criteria, will be asked to participate in the study. The aim is to enroll 40 subjects that will complete the whole study.

Recruited subjects will go through screening tests and if eligible, will undergo, within 18 days of screening, CT Guided chest PNB or FNA utilizing the ActiSight Needle Guidance system. Subjects will be observed and tested for at least an hour after the procedure to detect any serious complications. A follow-up will be conducted within 7-10 days after the procedure day for safety evaluations. Safety and accuracy data from all stages of the study will be collected and analyzed.

The effectiveness of the guidance system will be measured primarily by the frequency of reaching the intended targets, as determined by a final CT scan. Other measures will include the number of needle punctures and the number of intermediate CT scans needed to complete the procedure. The safety of the system will be measured by the frequency and severity of adverse events.

Procedure description:

First, a single-use, disposable pad (ActiSticker) is attached to the patient's skin over the point of needle insertion as selected by the interventionist. The pad incorporates reference objects that are easily detectable both on CT images and visually. A volume CT scan, covering at least the pad, the target lesion and adjacent structures is then performed. Next, the CT images from the volume scan are transferred to the ActiSight computer where the operator marks the target of the procedure, as well as all the reference points on the ActiSticker. Next, an optical sensor, also single-use and disposable, is attached to the top of the needle. By optically detecting all the reference points and relating them to their known positions on the CT images, the system can calculate the position of the top and the tip of the needle with relation to the target lesion. During the procedure, the system shows the user, on a graphic computer display, whether the needle is aimed directly at the target and how far the tip of the needle is from the intended target to help the user aim the insertion and guidance of the needle to the target.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18 years of age or older at the time of enrollment
* Subjects meeting all medical conditions for percutaneous chest aspiration/biopsy with safe path to lesion between ribs, however, not in the breast area in women or men with gynecomastia
* Single target pulmonary lesion greater than 10 mm in size (diameter) and depth of lesion greater than 40 mm from the skin
* Written informed consent to participate in the study
* Ability to comply with the requirements of the study procedures

Exclusion Criteria:

* Fibrous tissue or cyst in access path (not including target lesion)
* Hemophilia, thrombocytopenia, coagulopathy, or other elevated risk for bleeding or abnormal clotting
* Use of ticlodipine or similar antithrombotic medication
* For subjects taking warfarin or other anticoagulant medication, INR >1.3
* Pulmonary hypertension, heart failure, renal failure, or blood dyscrasia
* Patient is unable to comply with requirements of the procedure, i.e. holding breath
* Participation in any prior investigational trial within 30 days of enrollment
* Any form of substance abuse (including drug or alcohol abuse), psychiatric disorder, or any chronic condition that could, in the opinion of the investigator, of interfering with the conduct of the study.
* Subjects who are uncooperative or cannot follow instructions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2008-01; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Frequency of target reached within a radius of 5 mm from the preplanned targeted point as measured on the final CT scan | Measure evaluated during entire course of study

SECONDARY OUTCOMES:
Number of punctures required to obtain sample | Measure evaluated during entire course of study
Number of intermediate CT scans required to obtain sample | During entire course of study
An adequate sample obtained during the procedure | during entire course of study

CONTACTS AND LOCATIONS:
Overall Officials: Narinder Paul, MD, Principal Investigator — University Health Network, Toronto General Hospital; Uri Shreter, Ph.D., Study Director — ActiViews Ltd.
Locations (1):
- University Health Network, Toronto General Hospital, Toronto, Ontario, Canada